CLINICAL TRIAL: NCT06060444
Title: Evaluating a Telemedicine Neurological Consult Program for Drug-Induced Movement Disorders Using the RE-AIM Framework
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: Neurocrine Biosciences (Industry)
Responsible Party: Principal Investigator, Emily Houston, Principal Investigator, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00001579
Record Dates: First submitted 2023-06-10; First posted 2023-09-29 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Drug-Induced Movement Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- In-Person (Other): Control group
  Interventions: Other: In-person Consult
- Telemedicine (Experimental)
  Interventions: Other: Telemedicine Consult

INTERVENTIONS:
Other: Telemedicine Consult — Neurological consultation completed remotely
  Arms: Telemedicine
Other: In-person Consult — Neurological consultation completed in-person
  Arms: In-Person

SUMMARY:
In this pilot study, the investigators will evaluate care delivery via telemedicine to individuals with drug-induced movement disorders (DIMDs). DIMDs can be disabling, and prevention is important; but these disorders are often under-reported, under-recognized and poorly managed. Interprofessional telemedicine for movement disorders is feasible and may provide similar care as in-person visits; however, the majority of studies to date have shown benefit in Parkinson's disease and further validation in other movement disorders is necessary.

In this randomized controlled trial the aim is to study the acceptability, feasibility, and patient and clinician outcomes when a neurological consultation is provided for patients with DIMDs either in-person or through telemedicine. The investigators will apply the evaluation framework RE-AIM (Reach and Effectiveness, Adoption, Implementation, and Maintenance) to comprehensively assess the factors that may impact study success and program implementation. Mixed methods will be implemented to gather outcome data from mental health clinicians that refer patients and the patient participants.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Willing and able to provide consent
* Willing to have their Mental Health Clinician (MHC) share sensitive clinical information with the Neurology team
* Able to travel to Neurology clinic
* Have connectivity to Zoom using wi-fi or cellular data, either at home or a comfortable and private setting (such as MHC office)

Exclusion Criteria:

* Currently hospitalized
* Neurologist determines patient requires care outside of the scope of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Effectiveness; Client Satisfaction Questionnaire-8 (CSQ-8) | 12 months
  How satisfied are patients with the program

SECONDARY OUTCOMES:
Effectiveness; PROMIS 29+2 V2.1 | 12 months
  What are the impacts on patient health status
Effectiveness; referral forms and visit notes | 12 months
  Was there concordance in diagnosis between the MHC and movement disorder specialist
Effectiveness; visit notes | 12 months
  Was there an impact on care plan
Effectiveness; MHC survey and Qualitative Interviews | 12 months
  Were the MHCs Satisfied with the program

OTHER OUTCOMES:
Reach | 12 months
  In this study, are we able to enroll a sample that is representative of the patient population that experiences DIMDs
Adoption | 12 months
  Are there factors that determine whether a clinician will initiate participation in this program
Implementation | 12 months
  What barriers exist that may determine the feasibility of the study and neurological consultation
Maintenance; MHC survey and qualitative interviews | 12 months
  Could a telemedicine program similar to the one we develop for this study become a part of the routine organizational practices

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No
Currently there is no plan to share individual participant data (IPD) with other researchers.